CLINICAL TRIAL: NCT04638894
Title: Are Patient Characteristics and Treatment Characteristics Related to the Value of the Adult Spinal Deformity (ASD) Care Pathway in University Hospitals Leuven?
Brief Title: Variability in ASD (Adult Spinal Deformity) Value
Acronym: VIAV
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S63875
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Hospital Costs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Surgical treatment of patients with adult spinal deformity — Including all surgical interventions for patients with adult spinal deformity.

SUMMARY:
The study will examine if variability in created value (outcome/costs) over the care cycle for ASD patients can be explained by patient and treatment characteristics.

DETAILED DESCRIPTION:
Due to budget restrictions in health care, cost is a major challenge, particularly in chronic disorders affecting the ageing population for which advanced but often expensive medical technologies offer benefit. Stakeholders strive to define, assess and improve the so-called "value in healthcare" to achieve the best outcome at the lowest cost of care.

First and foremost, the investigator will try to examine if we can explain variability in the created value over the care cycle by patient and treatment characteristics. This knowledge can be used to optimize the value for the patients. Also, the investigator will try to compare the psychometric properties between the different versions of value equations, resulting from the use of different outcome tools to measure value.

Adult Spinal Deformity patients can take part in the study. This will be decided by clinical examination and radiographic evaluation and is based on at least one of the following criteria: 1) Coronal spinal curvature ≥20°, 2)Sagittal vertical axis (SVA) >5 cm, 3) Pelvic tilt >25°, 4) Thoracic kyphosis >60°. The patients have to be older than or equal to 18 years old at the time of surgery.

In line with the standard of care, the patients will be seen after 3 months, 6 months, 1 year and 2 years postoperatively. Pre- and post-operatively, questionnaires will be completed by the patients. The patient questionnaires EuroQol 5D (EQ-5D-3L and EQ-5D-5L) , Scoliosis Research Society 22 score (SRS-22), Oswestry disability Index, Core Outcome Measures Index score (COMI) and Work status will be completed by the patients during the baseline visit and on each follow-up moment at 3 months, 6 months, 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult Spinal Deformity patients
* Index Surgery from 15/03/2020 and 15/03/2022
* Age of 18 years old or older at the moment of the index surgery
* Patients treated in University Hospitals Leuven
* Patient has full understanding and is willing to participate (Informed consent)

Exclusion Criteria:

* • Patients younger than 18 years old at the moment of index surgery

  * Patients with an index surgery before 15/03/2020
  * Patients treated in other centers outside of University Hospitals Leuven

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of patients, diagnosed with ASD, with an index surgery between 15 march 2020 and 15 march 2022 at University Hospitals Leuven.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Generic Value | 2 years
  Generic outcome, measured via the EuroQol 5D (EQ-5D), divided by costs
Disease specific value: Scoliosis Research Society Outcomes Questionnaire (SRS-22) | 2 years
  Disease-specific value, measured via the Scoliosis Research Society Outcomes Questionnaire (SRS-22), divided by costs
Disease specific value: Oswestry Low Back Pain Disability Questionnaire (ODI) | 2 years
  Disease-specific value, measured via the Oswestry Low Back Pain Disability Questionnaire (ODI), divided by costs
Disease specific value: Core Outcome Measures Index (COMI) | 2 years
  Disease-specific value, measured via the Core Outcome Measures Index (COMI), divided by costs

SECONDARY OUTCOMES:
Workstatus | 2 years
  Workstatus, following the International Consortium for Health Outcomes Measurement (ICHOM) standard low back pain
Return to work | 2 years
  Return to work, following the International Consortium for Health Outcomes Measurement (ICHOM) standard low back pain

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Moke, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided